CLINICAL TRIAL: NCT06305715
Title: Radiation Prior to TKI to Delay Progression in Advanced Driver-Mutated Non-small Cell Lung Cancers (RadiaNCe Lung X)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jonathan Thompson, MD, MS, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00051658
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non-small cell lung cancer; radiation therapy; tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation therapy followed by mutation-matched TKI treatment (Experimental): Part 1 will enroll subjects who will be given radiation doses at the discretion of the treating physicians. Subjects with actionable driver mutation will continue to Part 2 and receive a standard-of-care TKI at the discretion of the treating oncologist.
  Interventions: Device: Radiation Therapy; Drug: Targeted TKI therapy

INTERVENTIONS:
Device: Radiation Therapy — Enrolled subjects will be given radiation doses, at the discretion of the treating physicians, that range from 24-60 Gy in 1-15 fractions with a minimum biologically effective dose (BED^10) of 58 Gy.
Drug: Targeted TKI therapy — Immediately following radiation therapy, subjects with an actionable driver mutation will receive a standard-of-care TKI. The choice of TKI will be at the discretion of the treating oncologist.

SUMMARY:
This prospective, two-part, single-arm, phase II trial is designed to evaluate whether the use of definitive radiation to the primary lung lesion prolongs progression-free survival (PFS) in treatment-naïve, metastatic, driver-mutated non-small cell lung cancers (NSCLC) patients who are subsequently placed on a tyrosine kinase inhibitor (TKI).

DETAILED DESCRIPTION:
This is a prospective, two-part, single-arm, phase II trial that will evaluate whether the use of definitive radiation to the primary lung lesion prolongs PFS in treatment-naïve, metastatic, driver-mutated NSCLC patients who are subsequently put on a TKI. Part 1 will enroll up to 34 patients who are are treatment-naïve and have metastatic NSCLC. Enrolled subjects will be given radiation doses, at the discretion of the treating physicians, that range from 24-60 Gy in 1-15 fractions with a minimum biologically effective dose (BED10) of 58 Gy.

Immediately following the completion of radiation therapy, patients who have an actionable driver mutation will be eligible to continue on to Part 2 of the study; those who do not meet the eligibility criteria for Part 2 will discontinue trial participation. Twenty-nine subjects will receive a standard-of-care targeted TKI therapy. The choice of TKI will be at the discretion of the treating oncologist, provided that their decision aligns with preferred TKIs per National Comprehensive Cancer Network (NCCN) guidelines. While on TKI therapy, patients will be assessed every three months for disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and survival.

ELIGIBILITY:
Inclusion Criteria Part 1

1. Age ≥18 years.
2. Patient must have a pathologically-confirmed diagnosis of non-small cell lung cancer (NSCLC).
3. An identifiable primary lung lesion must be present based on the consensus opinion of the medical oncology and radiation oncology investigators.
4. Patient did not previously receive radiation therapy to the primary lung lesion. Previous or concurrent palliative radiation to symptomatic metastatic lesions and definitive radiation to central nervous system metastases are allowable.
5. Patient must have advanced disease, either stage IV or stage IIIB/C that is not amenable to definitive multi-modality therapy.
6. Patient must not have received prior targeted therapy for NSCLC. A subject may receive up to 2 cycles of standard cytotoxic chemotherapy for NSCLC prior to trial enrollment. For example, a cycle of carboplatin and pemetrexed is given once every 3 weeks.
7. Patient must have measurable disease as defined by RECIST v1.1.
8. Patient must have Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 2.
9. Ability to understand a written informed consent document, and the willingness to sign it.

Inclusion Criteria Part 2

1. Must have an actionable driver mutation for which an Food and Drug Administration (FDA) -approved and/or National Comprehensive Cancer Network (NCCN) -recommended front-line TKI is available.

Exclusion Criteria:

1. Anticipated prognosis < 3 months.
2. Inability to swallow oral medications or history of GI abnormality that would impair absorption of oral medications.
3. Patients with prior or concurrent malignancy are eligible provided the investigator assesses this malignancy does not have potential to interfere with evaluation of the safety or efficacy of the study treatments.
4. Patient must not have any unresolved toxicities from prior cancer therapy greater than CTCAE grade 2 at time of study enrollment. Any grade alopecia is allowable.
5. Patient must not have medical contraindications, as determined by treating radiation oncologist, that would preclude safe delivery of radiation therapy.
6. Women must not be pregnant or breast-feeding. All females of childbearing potential must have negative blood or urine pregnancy testing within 14 days of study enrollment.
7. Women of childbearing potential and sexually active males must use effective methods of contraception for 14 days prior to study enrollment, while on study treatment, and for 4 months after the last targeted therapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Start of TKI treatment to 18 months
  The number of subjects without tumor progression based on RECIST v1.1 or death, whichever comes first. This will be measured from the start of TKI treatment until 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Thompson, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No